CLINICAL TRIAL: NCT01845805
Title: A Phase II Trial to Improve Outcomes in Patients With Resected Pancreatic Adenocarcinoma at High Risk for Recurrence Using Epigenetic Therapy
Brief Title: Trial to Improve Outcomes in Patients With Resected Pancreatic Cancer (Azacitidine)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J12138; NA_00076474 (Other: JHM IRB)
Record Dates: First submitted 2013-04-16; First posted 2013-05-03 (Estimated); Results first posted 2022-07-22 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Azacitidine; cc-486; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: CC-486 (Experimental): CC-486 (oral azacitidine), 300 mg total, taken daily on days 1-21 (of a 28 day cycle) for up to 12 cycles. Upon disease recurrence, subjects will start on a first-line chemotherapy.
  Interventions: Drug: oral azacitidine
- Arm B: observation (Active Comparator): Observation until disease recurrence. Upon disease recurrence, subjects will start on a first-line chemotherapy.
  Interventions: Other: Observation

INTERVENTIONS:
Drug: oral azacitidine
  Other Names: CC-486
  Arms: Arm A: CC-486
Other: Observation
  Arms: Arm B: observation

SUMMARY:
To improve progression free survival in high risk patients with resected pancreatic adenocarcinoma who have node positive disease, margin positive disease, and/or elevation in CA 19-9 treated with CC-486 (oral azacitidine) as compared to observation after completion of adjuvant therapy.

DETAILED DESCRIPTION:
This trial is for patients with resected pancreatic adenocarcinoma who have concluded adjuvant therapy or were deemed unable to receive adjuvant therapy with an elevated CA19-9 or node positive or margin positive disease. CA 19-9 elevation is defined as two levels > the institutional upper limit of normal (ULN) taken at least 2 weeks apart. These levels should be measured after adjuvant therapy has concluded or upon the decision that adjuvant therapy will not be offered. Patients will be randomized to one of two arms. Subjects enrolled due to node positive disease or R1 resection must be able to undergo randomization within 3 months of finishing adjuvant therapy or the decision that they are unable to take adjuvant therapy. Patients enrolling due to CA19-9 elevation can enroll any time after adjuvant therapy has completed. Arm A, the treatment arm, will be started on CC-486. Arm B, the control arm, will receive no additional therapy. In both arms, CA19-9 will be followed and CT scans (or MRI, if clinically indicated) will be done every three months. When patients have visible disease recurrence on imaging, CC-486 will be stopped and both groups will start first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age greater than or 18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Subjects must have a histologically confirmed pancreatic adenocarcinoma that has had an R0 (negative margins) or R1 (microscopically positive margins) resection.
* Subjects must have finished adjuvant therapy, which can include chemotherapy and/or chemoradiation therapy or have been determined to be unable to take adjuvant therapy. Although patients will be expected to complete chemoradiation or chemotherapy per physician recommendations, patients who are unable to complete chemotherapy ± radiation therapy secondary to dose limiting toxicities will be eligible provided they meet study criteria.
* Subjects enrolled due to node + disease or R1 resection must be able to undergo randomization within 3 months of finishing adjuvant therapy or the decision that they are unable to take adjuvant therapy. Patients enrolling due to CA 19-9 elevations can enroll any time after adjuvant therapy has completed.
* All previous cancer therapy including radiation, chemotherapy, and surgery, must have been discontinued at least 4 weeks prior to treatment in this study
* Subjects must either have a CA 19-9 value > the institutional ULN on two separate checks at least 2 weeks apart OR have had an R1 resection margin OR N1 nodal disease regardless of CA 19-9 level
* Subjects must be free of visible disease on imaging (CT, PETCT or MRI) evaluating chest, abdomen, and pelvis within 28 days of enrollment on the study.
* Life expectancy of greater than 12 weeks
* ECOG performance status of less than or equal to 1 at study entry
* Subjects must have normal organ and marrow function
* Free of prior malignancies for greater than or equal to 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast.
* Women of childbearing potential should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment with CC-486 or nab-paclitaxel. All men and women of childbearing potential must use effective methods of birth control throughout the study and for three months after completing treatment.
* Women of childbearing potential must have a negative serum or urine β-hCG pregnancy test at screening.
* Subjects must have < Grade 2 pre-existing peripheral neuropathy (per CTCAE)

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breastfeeding women.
* Use of any other chemotherapy, radiotherapy, or experimental drug or therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to enrollment on study or those who have not recovered from adverse events ≥ grade 1 due to agents administered more than 4 weeks earlier except for stable grade 2 neuropathy.
* Subjects may not receive any other concomitant investigational agents.
* Known or suspected hypersensitivity to 5-azacitidine or mannitol
* Known positive for HIV or infectious hepatitis, type B or C. HIV patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any known gastrointestinal disorders which would preclude oral administration of 5-azacitidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (4):
- United States (4):
  - Johns Hopkins, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Heumann TR, Baretti M, Sugar EA, Durham JN, Linden S, Lopez-Vidal TY, Leatherman J, Cope L, Sharma A, Weekes CD, O'Dwyer PJ, Reiss KA, Monga DK, Ahuja N, Azad NS. A randomized, phase II trial of oral azacitidine (CC-486) in patients with resected pancreatic adenocarcinoma at high risk for recurrence. Clin Epigenetics. 2022 Dec 3;14(1):166. doi: 10.1186/s13148-022-01367-8. PMID 36463226

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: CC-486 | Arm B: Observation
Started | 24 | 25
Completed | 6 | 9
Not Completed | 18 | 16
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Disease Progression | 13 | 14
Not completed — Drug-related Toxicity | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: CC-486 | Arm B: Observation | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 14 | 25
  >=65 years | 13 | 11 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 11 | 15 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 25 | 48
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 24 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression free survival is defined as the time from randomization until visible recurrence on any imaging modality, a confirmed biopsy, or death. Individuals lost to follow-up prior to having an event will be censored at the time of the last scan or biopsy.
Time Frame: 25 months
Population: Only 23/24 were evaluable for this outcome in Arm A
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: CC-486 | Arm B: Observation
Number analyzed (Participants) | 23 | 25
months | 9.2 [4.1 to 20.9] | 8.9 [3.4 to 24.6]

2. Secondary Outcome: Response Rate as Assessed by Number of Participants With Partial or Complete Response
Description: Response rate (partial response or complete response) to first-line chemotherapy when given after visible disease recurrence in patients primed with CC-486 compared to observation. Partial and complete responses were assessed by standard of care radiology reads and documented scan interpretations.
Time Frame: 11 months
Population: Evaluable participants for this outcome include participants with recurrence post-treatment with CC-486 who went on to receive first line chemotherapy and completed a follow-up scan that was available for review. Only 13/24 in Arm A and 13/25 in Arm B were evaluable for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: CC-486 | Arm B: Observation
Number analyzed (Participants) | 13 | 13
Participants | 1 | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization until death. Individuals lost to follow-up prior to death will be censored at the time of last physician contact.
Time Frame: 47 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: CC-486 | Arm B: Observation
Number analyzed (Participants) | 24 | 25
months | 33.8 [12.8 to 47.6] | 26.4 [17.8 to 46.7]

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were evaluated over 12 months. All-cause mortality was evaluated for up to 47 months.
Description: Only 23/24 participants in Arm A were assessed for Serious and Other (Not Including Serious) Adverse Events. Arm B (Observation) patients did not receive any treatment; therefore Serious and Other (Not Including Serious) Adverse Events were not collected. During the survival follow-up portion of the trial, patients in both Arms A and B were evaluated for all-cause mortality past the 12 month time frame of treatment and the assessment of adverse events.
Arm/Group | Arm A: CC-486 | Arm B: Observation
All-Cause Mortality (participants affected / at risk) | 15/24 | 14/25
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/0
Other Adverse Events (participants affected / at risk) | 23/23 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: CC-486 (N=23) | Arm B: Observation (N=0)
Weight Loss (Investigations) | 5 (5) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 14 (19) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 10 (15) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (21) | 0 (0)
Vomting (Gastrointestinal disorders) | 3 (4) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 5 (7) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (7) | 0 (0)
Anorexia (Gastrointestinal disorders) | 7 (7) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Oral abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 3 (3) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) — and administration site conditions
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (3) | 0 (0)
White blood cell count decreased (Investigations) | 6 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT01845805/Prot_SAP_000.pdf